CLINICAL TRIAL: NCT02792192
Title: A Phase Ib/II, Open-Label Study of the Safety and Pharmacology of Atezolizumab Administered With or Without Bacille Calmette-Guérin in Patients With High-Risk Non-Muscle-Invasive Bladder Cancer
Brief Title: Safety and Pharmacology Study of Atezolizumab Alone and in Combination With Bacille Calmette-Guérin (BCG) in High-Risk Non-Muscle-Invasive Bladder Cancer (NMIBC) Participants
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early as the study had met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO29635
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab; BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) (Experimental): Participants will receive atezolizumab 1200 mg IV infusion q3w, for a maximum of 32 doses or 96 weeks of therapy, whichever comes first.
  Interventions: Drug: Atezolizumab
- Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) (Experimental): During BCG induction course (12 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of six doses. During BCG maintenance course 1 (12 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of three doses. Optional BCG maintenance courses 2-5 (each 24 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of eight doses per course plus BCG at the assigned dose weekly for a total of three doses per course.
  Interventions: Drug: Atezolizumab; Biological: Bacille Calmette-Guérin
- Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) (Experimental): During BCG induction course (12 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of six doses. During BCG maintenance course 1 (12 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of three doses. During BCG maintenance courses 2-5 (each 24 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of eight doses per course plus BCG at the assigned dose weekly for a total of three doses per course.
  Interventions: Drug: Atezolizumab; Biological: Bacille Calmette-Guérin
- Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC) (Experimental): During BCG induction course (12 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of six doses. During BCG maintenance course 1 (12 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of three doses. During BCG maintenance courses 2-5 (each 24 weeks), participants will receive atezolizumab 1200 mg IV infusion q3w for a total of eight doses per course plus BCG at the assigned dose weekly for a total of three doses per course.
  Interventions: Drug: Atezolizumab; Biological: Bacille Calmette-Guérin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as per the schedule specified in respective arm.
  Other Names: MPDL3280A
Biological: Bacille Calmette-Guérin — For Cohort 1B, BCG will be administered (intravesically) at de-escalated doses. De-escalation will be allowed for up to three dose levels of BCG: full dose (50 mg), 66% of full dose, and 33% of full dose. After the MTD or MAD is determined for Cohort 1B, MTD/MAD will be used for all subsequent participants enrolled into Cohorts 1B, 2, and 3 (provided MAD or MTD is determined to be either full dose or 66% of a full BCG dose).
  Other Names: OncoTICE®
  Arms: Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC); Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC); Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)

SUMMARY:
This Phase Ib/II study is designed to assess the safety, tolerability, pharmacokinetics, immunogenicity, patient reported outcomes (PROs), and preliminary anti-tumor activity of atezolizumab administered by intravenous (IV) infusion alone and in combination with intravesical BCG in high-risk NMIBC participants. The study will be conducted in following cohorts: Cohort 1A, Cohort 1B, Cohort 2, and Cohort 3. Atezolizumab will be administered at a fixed dose of 1200 milligrams (mg) every 3 weeks (q3w) for a maximum of 96 weeks. BCG will be administered to evaluate dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), or maximum administered dose (MAD). De-escalation will be allowed for up to three dose levels of BCG (full dose [50 mg], 66 percent [%] of a full dose, and 33% of a full dose [Cohort 1B only]). After the MTD or MAD is determined for Cohort 1B, this dose will be used for all subsequent participants enrolled into Cohorts 1B, 2, and 3, unless the MTD is determined to be 33% of a full BCG dose. If MTD is determined to be 33% of a full BCG dose, then, no participants will be enrolled into Cohorts 2 and 3 until an assessment of the safety and activity of the combination of atezolizumab plus 33% of a full BCG dose is completed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-muscle-invasive transitional cell carcinoma (TCC) of the bladder with carcinoma in-situ (CIS)
* High-risk NMIBC defined by the following:

BCG-unresponsive NMIBC:

Persistence of high-grade CIS at 6 months following an adequate course of BCG; or Stage/grade progression at 3 months after induction BCG; or Recurrence of high-grade CIS after achieving a disease-free state (i.e., CR) following induction of an adequate course of BCG that occurs less than (<) 6 months after the last exposure to BCG

BCG-relapsing NMIBC:

Recurrence of high-grade CIS after achieving a disease-free state following induction of an adequate course of BCG that occurs greater than or equal to (>/=) 6 months after the last exposure to BCG

Very high-risk (VHR) BCG-naïve NMIBC:

VHR NMIBC, defined as having at least 1 of the following: Multiple and/or large (greater than [>] 3 centimeters [cm]) T1, (HG/G3) tumors; T1, (HG/G3) tumor with concurrent CIS; T1, G3 with CIS in prostatic urethra; Micropapillary variant of non-muscle invasive urothelial carcinoma

* For BCG-unresponsive and BCG-relapsing NMIBC, participants must have received an adequate course of BCG
* Resection of all pTa/pT1 papillary disease
* No prior radiation to bladder or pelvic region
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to (</=) 2;
* Life expectancy >/=12 weeks
* Adequate hematologic and end-organ function
* Creatinine clearance >/=30 milliliters per minute (mL/min) (calculated using the Cockcroft-Gault formula)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 5 months after the last dose of study drug. Women must refrain from donating eggs during this same period.
* For men receiving BCG: Agreement to remain abstinent (refrain from sexual intercourse) or use a condom
* Tumor tissue biopsy within 60 days prior to study entry or availability of an archival specimen obtained within 60 days of study screening

Exclusion Criteria:

* Evidence of locally advanced, metastatic, muscle-invasive, and/or extravesical bladder cancer
* Any malignancy within 5 years prior to Cycle 1, Day 1
* History of autoimmune disease, idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or active pneumonitis
* Signs or symptoms of infection within 2 weeks prior to the first dose of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to the first dose of study treatment
* Treatment with any approved anti-cancer therapy within 3 weeks prior to the first dose of study treatment
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 4 weeks prior to the first dose of study treatment
* Pregnant or lactating women, or women intending to become pregnant during the study
* Prior allogeneic stem cell or solid organ transplantation
* Positive test for human immunodeficiency virus (HIV)
* Active hepatitis B or C and/or tuberculosis
* Severe infections within 28 days prior to the first dose of study treatment
* Significant cardiovascular disease
* Major surgical procedure other than for diagnosis within 4 weeks prior to the first dose of study treatment, or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live/attenuated vaccine within 4 weeks prior to the first dose of study treatment, within 5 months following the administration of the last dose of study drug, or anticipation that such a live/attenuated vaccine will be required during the study
* History of prior significant toxicity or intolerance to BCG requiring discontinuation of treatment
* History of prior systemic BCG infection
* History of immunosuppression, or conditions associated with congenital or acquired immune deficiency
* Concurrent febrile illness, urinary tract infection, or gross hematuria
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies
* Treatment with systemic immunostimulatory agents within 6 weeks or five half-lives of the drug, whichever is shorter, prior to the first dose of study treatment
* Treatment with systemic immunosuppressive medications within 2 weeks prior to the first dose of study treatment, or anticipated requirement for systemic immunosuppressive medications during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - Stanford Univ., Stanford, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins Kimmel Cancer Center, Office of Research Administration, Baltimore, Maryland
  - The Montefiore Medical Center & The Albert Einstein College of Medicine; Department of Urology, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - VA Portland Healthcare System, Portland, Oregon

REFERENCES:
- [Derived] Inman BA, Hahn NM, Stratton K, Kopp R, Sankin A, Skinner E, Pohar K, Gartrell BA, Pham S, Rishipathak D, Mariathasan S, Davarpanah N, Carter C, Steinberg GD. A Phase 1b/2 Study of Atezolizumab with or Without Bacille Calmette-Guerin in Patients with High-risk Non-muscle-invasive Bladder Cancer. Eur Urol Oncol. 2023 Jun;6(3):313-320. doi: 10.1016/j.euo.2023.01.013. Epub 2023 Feb 15. PMID 36803840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled only in Cohort 1 of this study. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1 (BCG-unresponsive cohort), as the study had met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Groups:
- Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC): Participants received atezolizumab 1200 mg IV infusion q3w, for a maximum of 32 doses or 96 weeks of therapy, whichever comes first.
- Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC): During BCG induction course (12 weeks), participants received atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of six doses. During BCG maintenance course 1 (12 weeks), participants received atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of three doses. Optional BCG maintenance courses 2-5 (each 24 weeks), participants received atezolizumab 1200 mg IV infusion q3w for a total of eight doses per course plus BCG at the assigned dose weekly for a total of three doses per course.
- Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC); Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC): During BCG induction course (12 weeks), participants were to receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of six doses. During BCG maintenance course 1 (12 weeks), participants were to receive atezolizumab 1200 mg IV infusion q3w for a total of four doses plus BCG at the assigned dose weekly for a total of three doses. During BCG maintenance courses 2-5 (each 24 weeks), participants were to receive atezolizumab 1200 mg IV infusion q3w for a total of eight doses per course plus BCG at the assigned dose weekly for a total of three doses per course.
Period: Overall Study
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Started | 12 | 12 | 0 | 0
Completed | 0 | 1 | 0 | 0
Not Completed | 12 | 11 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Informed Consent Withdrawn | 4 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0
Not completed — Study Terminated By Sponsor | 6 | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were enrolled only in Cohort 1 of this study. The Sponsor decided to stop further enrollment for Cohorts 2 and 3 after the enrollment of 24 participants in Cohort 1 (BCG-unresponsive cohort), as the study had met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC) | Total
Number analyzed (Participants) | 12 | 12 | 0 | 0 | 24
Age, Continuous [Mean (Standard Deviation); unit: Year] | 72.7 (13.2) | 72.1 (9.0) |  |  | 72.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 |  |  | 2
  Male | 12 | 10 |  |  | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 12 | 11 | 0 | 0 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 0 | 4
  White | 8 | 10 | 0 | 0 | 18
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with at least one adverse event during the study.
Time Frame: From Baseline up to end of study (up to approximately 4.3 years)
Population: All participants were included in the safety-evaluable population, defined as all participants treated with any amount of study drug. Participants were enrolled only in Cohort 1 of this study. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 12 | 12 | 0 | 0
Percentage of participants | 100 | 100 |  |

2. Primary Outcome: Cohort 1B: Percentage of Participants With DLTs of BCG
Description: Percentage of participants with dose-limiting toxicities (DLT) of BCG in Cohort 1B.
Time Frame: Days 1-21
Population: All participants were included in the safety-evaluable population, defined as all participants treated with any amount of study drug. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC)
Number analyzed (Participants) | 12
Percentage of participants | 16.7

3. Primary Outcome: Cohort 1B: MAD of BCG
Description: Maximum administered dose (MAD) of BCG.
Time Frame: Days 1-21
Population: as for outcome 2
Measure: Number; unit: mg
Arm/Group | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC)
Number analyzed (Participants) | 12
mg | 50

4. Primary Outcome: Percentage of Participants With Complete Response (CR) as Assessed by the Investigator on the Basis of Cystoscopy and Urine Cytology at Month 6
Description: CR at 6 months after the start of study treatment as assessed by the investigator on the basis of cystoscopic assessment and urine cytology.
Time Frame: 6 months
Population: Efficacy evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 12 | 12 | 0 | 0
Percentage of participants | 33.3 [9.9 to 65.1] | 41.7 [15.2 to 72.3] |  |

5. Secondary Outcome: Percentage of Participants With CR as Assessed by the Investigator on the Basis of Cystoscopy and Urine Cytology at Month 3
Description: CR at the 3-month disease assessment, evaluated by both cystoscopy and cytology.
Time Frame: 3 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 12 | 12 | 0 | 0
Percentage of participants | 16.7 [2.1 to 48.4] | 41.7 [15.2 to 72.3] |  |

6. Secondary Outcome: Duration of CR, as Assessed on the Basis of Cystoscopy and Urine Cytology
Description: Duration of CR will be defined for participants with a CR as the time from the first occurrence of a documented complete response to recurrence of high-grade NMIBC or death from any cause.
Time Frame: From first occurence of a documented CR until the time of recurrence of NMIBC or death from any cause (up to approximately 4.3 years)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 4 | 5 | 0 | 0
Months
  Participants With CR at 6 Months | 6.80 [3.06 to NA] — Upper limit not estimable. Range: 3.06 to 22.3* months. * Indicating a censored observation for CR ongoing at last follow-up. | NA [NA to NA] — Median duration of CR was not reached. No participants had a recurrence event. |  |
  Participants With CR at 3 Months: number analyzed (Participants) | 2 | 5 | 0 | 0
  Participants With CR at 3 Months | NA [NA to NA] — Median duration of CR was not reached. For these 2 patients, CR was ongoing with duration of CR 3.61* and 22.3* months. | NA [3.71 to NA] — Median duration of CR was not reached. One patient had a recurrence event (duration of CR 3.71 months). For the remaining 4 patients, CR was ongoing with duration of CR ranging from 2.89* to 24.5* months. |  |

7. Secondary Outcome: Percentage of Participants With Recurrence-Free Survival (RFS), as Assessed on the Basis of Cystoscopy and Urine Cytology
Description: RFS rate at 6, 12, and 18 months, defined as the proportion of patients who are alive and free of persistent/recurrent high-grade NMIBC.
Time Frame: 6, 12 and 18 months
Population: Efficacy evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC. Data for RFS was not collected as the study was stopped early.
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Bladder-Intact Disease-Free Survival (DFS), as Assessed on the Basis of Cystoscopy and Urine Cytology
Description: Bladder-intact DFS was defined as the time from the first study treatment to earliest evidence of progression to muscle-invasive disease in the bladder, regional pelvic progression, distant metastasis, bladder cancer-related death, or cystectomy.
Time Frame: From first study treatment to earliest evidence of progression to muscle-invasive disease in the bladder, regional pelvic progression, distant metastasis, bladder cancer-related death, or cystectomy or death from any cause (up to approximately 4.3 years)
Population: Efficacy evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC. Data for DFS was not collected as the study was stopped early.
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Progression-Free Survival (PFS), as Assessed on the Basis of Cystoscopy and Urine Cytology
Description: PFS, defined as the time from the first study treatment to the first occurrence of progression to muscle-invasive disease based on cystoscopy and urine cytology or death from any cause.
Time Frame: Time from first study treatment to the first occurrence of progression to muscle-invasive disease or death from any cause (up to approximately 4.3 years)
Population: Efficacy evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC. Data for PFS was not collected as the study was stopped early.
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Cystectomy-Free Survival (CFS), as Assessed on the Basis of Cystoscopy and Urine Cytology
Description: Cystectomy-free survival, defined as from start of study treatment to bladder removal for any cause or death from any cause.
Time Frame: Time from first study treatment to cystectomy or death from any cause (up to approximately 4.3 years)
Population: Efficacy evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC. Data for CFS was not collected as the study was stopped early.
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Overall Survival
Time Frame: Time from first study treatment to death from any cause (up to approximately 4.3 years)
Population: Efficacy evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1), as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC. Data for OS was not collected as the study was stopped early.
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Maximum Observed Serum Concentration of Atezolizumab (Cmax)
Description: Maximum observed serum concentration of Atezolizumab (Cmax)
Time Frame: Cycle 1 Day 1 post-dose (Cycle length=21 days)
Population: PK evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 12 | 11 | 0 | 0
μg/mL | 413 (109) | 310 (63.7) |  |

13. Secondary Outcome: Minimum Observed Serum Concentration of Atezolizumab (Cmin)
Description: Minimum observed serum concentration of atezolizumab (Cmin)
Time Frame: Pre-dose (0 hr) on Day 1 of Cycles 2, 3, 4 and 8 (Cycle length=21 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 12 | 12 | 0 | 0
μg/mL
  Cycle 2 Day 1: number analyzed (Participants) | 12 | 10 | 0 | 0
  Cycle 2 Day 1 | 92.2 (14.9) | 90.5 (42.6) |  |
  Cycle 3 Day 1 | 143 (26.1) | 133 (74.4) |  |
  Cycle 4 Day 1: number analyzed (Participants) | 12 | 11 | 0 | 0
  Cycle 4 Day 1 | 174 (38.4) | 162 (91.1) |  |
  Cycle 8 Day 1: number analyzed (Participants) | 9 | 10 | 0 | 0
  Cycle 8 Day 1 | 211 (59.4) | 192 (117) |  |

14. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibody (ADA) Response to Atezolizumab
Description: Percentage of participants with anti-therapeutic antibody (ADA) response to atezolizumab.
Time Frame: Pre-dose (0 hr) on Day 1 of Cycles 1, 2, 3, 4, 8, 16, 24 (Cycle length=21 days), end of atezolizumab treatment (up to 96 weeks), 120 days after end of atezolizumab treatment (up to 113 weeks)
Population: ADA evaluable participants. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
Number analyzed (Participants) | 12 | 12 | 0 | 0
Percentage of participants
  Baseline prevalence: number analyzed (Participants) | 11 | 12 | 0 | 0
  Baseline prevalence | 9.1 | 0 |  |
  Post-Baseline Treatment-Emergent | 8.3 | 41.7 |  |

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 29 September 2020 (up to 4.3 years)
Description: The Safety Evaluable Population includes all participants treated with any amount of study drug (atezolizumab or BCG).
  Participants were enrolled only in Cohort 1 of this study. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1, as the study met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.
Arm/Group | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC)
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/12 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/12 | 3/12 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 11/12 | 12/12 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) (N=12) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) (N=12) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) (N=0) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC) (N=0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | NA | NA
Complication associated with device (General disorders) | 0 (0) | 1 (1) | NA | NA
Pyrexia (General disorders) | 1 (1) | 0 (0) | NA | NA
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | NA | NA
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A: Atezolizumab (BCG-unresponsive NMIBC) (N=12) | Cohort 1B: Atezolizumab + BCG (BCG-unresponsive NMIBC) (N=12) | Cohort 2: Atezolizumab + BCG (BCG-relapsing NMIBC) (N=0) | Cohort 3: Atezolizumab + BCG (BCG-naive NMIBC) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | NA | NA
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | NA | NA
Dry eye (Eye disorders) | 1 (1) | 0 (0) | NA | NA
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | NA | NA
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA | NA
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA | NA
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | NA | NA
Chills (General disorders) | 1 (1) | 0 (0) | NA | NA
Fatigue (General disorders) | 7 (9) | 2 (2) | NA | NA
Influenza like illness (General disorders) | 0 (0) | 2 (2) | NA | NA
Injury associated with device (General disorders) | 1 (1) | 0 (0) | NA | NA
Mucosal inflammation (General disorders) | 1 (2) | 0 (0) | NA | NA
Oedema (General disorders) | 0 (0) | 1 (1) | NA | NA
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | NA | NA
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | NA | NA
Pyrexia (General disorders) | 2 (2) | 1 (1) | NA | NA
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | NA | NA
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | NA | NA
Atypical mycobacterial pneumonia (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Cystitis (Infections and infestations) | 1 (2) | 0 (0) | NA | NA
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Influenza (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Pustule (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | NA | NA
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | NA | NA
Amylase increased (Investigations) | 0 (0) | 1 (1) | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (4) | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | NA | NA
Blood creatinine increased (Investigations) | 0 (0) | 2 (8) | NA | NA
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (5) | NA | NA
Platelet count decreased (Investigations) | 0 (0) | 1 (9) | NA | NA
Weight decreased (Investigations) | 1 (1) | 0 (0) | NA | NA
Weight increased (Investigations) | 0 (0) | 1 (2) | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | NA | NA
Anosmia (Nervous system disorders) | 0 (0) | 1 (1) | NA | NA
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | NA | NA
Headache (Nervous system disorders) | 1 (2) | 0 (0) | NA | NA
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | NA | NA
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | NA | NA
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | NA | NA
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | NA | NA
Bladder spasm (Renal and urinary disorders) | 1 (1) | 5 (5) | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (7) | NA | NA
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | NA | NA
Dysuria (Renal and urinary disorders) | 2 (2) | 4 (6) | NA | NA
Haematuria (Renal and urinary disorders) | 0 (0) | 5 (5) | NA | NA
Micturition urgency (Renal and urinary disorders) | 0 (0) | 2 (4) | NA | NA
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | NA | NA
Pollakiuria (Renal and urinary disorders) | 0 (0) | 6 (8) | NA | NA
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (2) | NA | NA
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | NA | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | NA | NA
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA | NA
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (3) | NA | NA
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA | NA
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | NA | NA
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | NA | NA

LIMITATIONS AND CAVEATS:
Participants were enrolled only in Cohort 1 of this study. The Sponsor decided not to enroll participants in Cohorts 2 and 3 after the enrollment of 24 patients in Cohort 1 (BCG-unresponsive cohort), as the study had met its goals of providing preliminary safety and efficacy information for atezolizumab monotherapy alone and in combination with BCG in NMIBC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02792192/Prot_SAP_000.pdf